CLINICAL TRIAL: NCT02173769
Title: AKTIV: Changes in Physical Functioning in Patients With COPD During Therapy With a Combination of Spiriva® Respimat® + Striverdi® Respimat® or Spiriva® 18 Mikrogramm + Striverdi® Respimat®
Brief Title: Changes in Physical Functioning in Patients With COPD During Therapy With a Combination Inhalation Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1222.56
Record Dates: First submitted 2014-06-24; First posted 2014-06-25 (Estimated); Results first posted 2016-04-01 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Adults with COPD
  Interventions: Drug: Spiriva® Respimat®; Drug: Striverdi® Respimat®

INTERVENTIONS:
Drug: Spiriva® Respimat® — Spiriva® Respimat® plus Striverdi® Respimat® or Spiriva® 18 Microgramm plus Striverdi® Respimat®
Drug: Striverdi® Respimat® — Spiriva® Respimat® plus Striverdi® Respimat® or Spiriva® 18 Microgramm plus Striverdi® Respimat®

SUMMARY:
The decrease in physical activity due to increasing dyspnoea that over time leads to a steadily worsening condition and increasing restriction of physical functioning is a key problem for COPD patients and affects even the early stages.

Clinical studies to investigate both Spiriva® and Striverdi® Respimat® have demonstrated a marked improvement in physical exercise capacity.

However, there have so far been no data from the daily practice setting about everyday functioning on combination treatment with Spiriva® Respimat® plus Striverdi® Respimat® or Spiriva® 18 Mikrogramm plus Striverdi® Respimat® in patients requiring treatment with 2 long-acting bronchodilators.

The objective of this NIS is to measure changes in physical functioning as a surrogate for physical activity and exercise capacity in COPD patients on treatment with Spiriva® Respimat® plus Striverdi® Respimat® or Spiriva® 18 Mikrogramm plus Striverdi® Respimat® in routine daily treatment (so-called real life setting).

ELIGIBILITY:
Inclusion criteria:

* Female and male patients >= 40 years
* COPD GOLD 2014 B - D
* Treatment with Spiriva® Respimat® plus Striverdi® Respimat® or Spiriva® 18 Microgramm plus Striverdi® Respimat® acc. to the Summary of Product Characteristics (SmPC), no change of routine diagnostics and treatment
* Signed informed consent form before inclusion into the non-interventional study (NIS)

Exclusion criteria:

* Patients with contraindications acc. to the Summary of Product Characteristics (SmPC)
* pregnant and breastfeeding women
* patients who are taking part in a different non-interventional study (NIS) or an interventional clinical study at the same time are not to be enrolled

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Probability Sample
Enrollment: 1845 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (701):
- Germany (701):
  - Boehringer Ingelheim Investigational Site 1, Aachen
  - Boehringer Ingelheim Investigational Site 2, Ahaus
  - Boehringer Ingelheim Investigational Site 3, Aichtal
  - Boehringer Ingelheim Investigational Site 4, Aldenhoven
  - Boehringer Ingelheim Investigational Site 5, Alfeld
  - Boehringer Ingelheim Investigational Site 6, Altötting
  - Boehringer Ingelheim Investigational Site 7, Ansbach
  - Boehringer Ingelheim Investigational Site 10, Asbach-Bäumenheim
  - Boehringer Ingelheim Investigational Site 8, Asbach-Bäumenheim
  - Boehringer Ingelheim Investigational Site 9, Asbach-Bäumenheim
  - Boehringer Ingelheim Investigational Site 12, Auerbach
  - Boehringer Ingelheim Investigational Site 13, Auerbach
  - Boehringer Ingelheim Investigational Site 14, Auerbach
  - Boehringer Ingelheim Investigational Site 15, Augsburg
  - Boehringer Ingelheim Investigational Site 16, Augsburg
  - Boehringer Ingelheim Investigational Site 11, Aßlar
  - Boehringer Ingelheim Investigational Site 17, Bacharach
  - Boehringer Ingelheim Investigational Site 18, Bad Friedrichshall
  - Boehringer Ingelheim Investigational Site 19, Bad Krozingen
  - Boehringer Ingelheim Investigational Site 20, Bad Langensalza
  - Boehringer Ingelheim Investigational Site 21, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site 22, Bad Lippspringe
  - Boehringer Ingelheim Investigational Site 23, Bad Reichenhall
  - Boehringer Ingelheim Investigational Site 24, Bad Sachsa
  - Boehringer Ingelheim Investigational Site 25, Bad Soden
  - Boehringer Ingelheim Investigational Site 26, Bad Soden-Salmünster
  - Boehringer Ingelheim Investigational Site 27, Bad Windsheim
  - Boehringer Ingelheim Investigational Site 28, Bad Wörishofen
  - Boehringer Ingelheim Investigational Site 29, Baden-Baden
  - Boehringer Ingelheim Investigational Site 30, Balingen
  - Boehringer Ingelheim Investigational Site 31, Beelitz-Heilstätten
  - Boehringer Ingelheim Investigational Site 32, Beelitz-Heilstätten
  - Boehringer Ingelheim Investigational Site 33, Bensheim
  - Boehringer Ingelheim Investigational Site 34, Bensheim
  - Boehringer Ingelheim Investigational Site 35, Berkatal-Frankershausen
  - Boehringer Ingelheim Investigational Site 36, Berlin
  - Boehringer Ingelheim Investigational Site 37, Berlin
  - Boehringer Ingelheim Investigational Site 38, Berlin
  - Boehringer Ingelheim Investigational Site 39, Berlin
  - Boehringer Ingelheim Investigational Site 40, Berlin
  - Boehringer Ingelheim Investigational Site 41, Berlin
  - Boehringer Ingelheim Investigational Site 42, Berlin
  - Boehringer Ingelheim Investigational Site 43, Berlin
  - Boehringer Ingelheim Investigational Site 44, Berlin
  - Boehringer Ingelheim Investigational Site 45, Berlin
  - Boehringer Ingelheim Investigational Site 46, Berlin
  - Boehringer Ingelheim Investigational Site 47, Berlin
  - Boehringer Ingelheim Investigational Site 48, Berlin
  - Boehringer Ingelheim Investigational Site 49, Berlin
  - Boehringer Ingelheim Investigational Site 50, Berlin
  - Boehringer Ingelheim Investigational Site 51, Berlin
  - Boehringer Ingelheim Investigational Site 52, Berlin
  - Boehringer Ingelheim Investigational Site 53, Berlin
  - Boehringer Ingelheim Investigational Site 54, Berlin
  - Boehringer Ingelheim Investigational Site 55, Berlin
  - Boehringer Ingelheim Investigational Site 56, Berlin
  - Boehringer Ingelheim Investigational Site 57, Berlin
  - Boehringer Ingelheim Investigational Site 58, Berlin
  - Boehringer Ingelheim Investigational Site 59, Berlin
  - Boehringer Ingelheim Investigational Site 60, Berlin
  - Boehringer Ingelheim Investigational Site 61, Berlin
  - Boehringer Ingelheim Investigational Site 64, Bernkastel
  - Boehringer Ingelheim Investigational Site 65, Biberach
  - Boehringer Ingelheim Investigational Site 66, Biberach
  - Boehringer Ingelheim Investigational Site 67, Biberach
  - Boehringer Ingelheim Investigational Site 68, Bielefeld
  - Boehringer Ingelheim Investigational Site 69, Bielefeld
  - Boehringer Ingelheim Investigational Site 70, Blankenheim
  - Boehringer Ingelheim Investigational Site 71, Bocholt
  - Boehringer Ingelheim Investigational Site 72, Bocholt
  - Boehringer Ingelheim Investigational Site 73, Bochum
  - Boehringer Ingelheim Investigational Site 74, Bockenheim
  - Boehringer Ingelheim Investigational Site 75, Bodenwerder
  - Boehringer Ingelheim Investigational Site 76, Bonn
  - Boehringer Ingelheim Investigational Site 77, Bonn
  - Boehringer Ingelheim Investigational Site 78, Bonn
  - Boehringer Ingelheim Investigational Site 79, Bonn
  - Boehringer Ingelheim Investigational Site 80, Bonn
  - Boehringer Ingelheim Investigational Site 81, Bottrop
  - Boehringer Ingelheim Investigational Site 82, Bottrop
  - Boehringer Ingelheim Investigational Site 83, Brandenburg
  - Boehringer Ingelheim Investigational Site 84, Braunschweig
  - Boehringer Ingelheim Investigational Site 85, Bremen
  - Boehringer Ingelheim Investigational Site 86, Bremen
  - Boehringer Ingelheim Investigational Site 87, Bremen
  - Boehringer Ingelheim Investigational Site 88, Bremen
  - Boehringer Ingelheim Investigational Site 89, Bremen
  - Boehringer Ingelheim Investigational Site 90, Bruchsal
  - Boehringer Ingelheim Investigational Site 91, Bruchweiler-Bärenbach
  - Boehringer Ingelheim Investigational Site 92, Buchbach
  - Boehringer Ingelheim Investigational Site 95, Burg
  - Boehringer Ingelheim Investigational Site 96, Burg
  - Boehringer Ingelheim Investigational Site 97, Burgheim
  - Boehringer Ingelheim Investigational Site 98, Burgstädt
  - Boehringer Ingelheim Investigational Site 93, Bünde
  - Boehringer Ingelheim Investigational Site 94, Bünde
  - Boehringer Ingelheim Investigational Site 100, Cham
  - Boehringer Ingelheim Investigational Site 101, Chemnitz
  - Boehringer Ingelheim Investigational Site 102, Chemnitz
  - Boehringer Ingelheim Investigational Site 103, Chemnitz
  - Boehringer Ingelheim Investigational Site 104, Claußnitz
  - Boehringer Ingelheim Investigational Site 105, Cloppenburg
  - Boehringer Ingelheim Investigational Site 106, Coburg
  - Boehringer Ingelheim Investigational Site 340, Cologne
  - Boehringer Ingelheim Investigational Site 341, Cologne
  - Boehringer Ingelheim Investigational Site 342, Cologne
  - Boehringer Ingelheim Investigational Site 343, Cologne
  - Boehringer Ingelheim Investigational Site 344, Cologne
  - Boehringer Ingelheim Investigational Site 345, Cologne
  - Boehringer Ingelheim Investigational Site 346, Cologne
  - Boehringer Ingelheim Investigational Site 347, Cologne
  - Boehringer Ingelheim Investigational Site 348, Cologne
  - Boehringer Ingelheim Investigational Site 349, Cologne
  - Boehringer Ingelheim Investigational Site 350, Cologne
  - Boehringer Ingelheim Investigational Site 351, Cologne
  - Boehringer Ingelheim Investigational Site 352, Cologne
  - Boehringer Ingelheim Investigational Site 353, Cologne
  - Boehringer Ingelheim Investigational Site 107, Cottbus
  - Boehringer Ingelheim Investigational Site 108, Cottbus
  - Boehringer Ingelheim Investigational Site 109, Cottbus
  - Boehringer Ingelheim Investigational Site 110, Cottbus
  - Boehringer Ingelheim Investigational Site 111, Cottbus
  - Boehringer Ingelheim Investigational Site 112, Cottbus
  - Boehringer Ingelheim Investigational Site 113, Cottbus
  - Boehringer Ingelheim Investigational Site 114, Cottbus
  - Boehringer Ingelheim Investigational Site 115, Darmstadt
  - Boehringer Ingelheim Investigational Site 116, Deggendorf
  - Boehringer Ingelheim Investigational Site 117, Delitzsch
  - Boehringer Ingelheim Investigational Site 118, Delitzsch
  - Boehringer Ingelheim Investigational Site 119, Dessau
  - Boehringer Ingelheim Investigational Site 120, Dessau
  - Boehringer Ingelheim Investigational Site 121, Dessau
  - Boehringer Ingelheim Investigational Site 122, Dortmund
  - Boehringer Ingelheim Investigational Site 123, Dortmund
  - Boehringer Ingelheim Investigational Site 124, Dortmund
  - Boehringer Ingelheim Investigational Site 125, Dortmund
  - Boehringer Ingelheim Investigational Site 126, Dortmund
  - Boehringer Ingelheim Investigational Site 127, Dortmund
  - Boehringer Ingelheim Investigational Site 128, Drensteinfurt
  - Boehringer Ingelheim Investigational Site 129, Dresden
  - Boehringer Ingelheim Investigational Site 130, Dudenhofen
  - Boehringer Ingelheim Investigational Site 131, Duisburg
  - Boehringer Ingelheim Investigational Site 132, Duisburg
  - Boehringer Ingelheim Investigational Site 133, Duisburg
  - Boehringer Ingelheim Investigational Site 134, Duisburg
  - Boehringer Ingelheim Investigational Site 135, Duisburg
  - Boehringer Ingelheim Investigational Site 136, Duisburg
  - Boehringer Ingelheim Investigational Site 137, Duisburg
  - Boehringer Ingelheim Investigational Site 138, Düsseldorf
  - Boehringer Ingelheim Investigational Site 139, Düsseldorf
  - Boehringer Ingelheim Investigational Site 140, Düsseldorf
  - Boehringer Ingelheim Investigational Site 141, Düsseldorf
  - Boehringer Ingelheim Investigational Site 142, Düsseldorf
  - Boehringer Ingelheim Investigational Site 143, Ehrenkirchen
  - Boehringer Ingelheim Investigational Site 144, Eisenach
  - Boehringer Ingelheim Investigational Site 145, Eisenhüttenstadt
  - Boehringer Ingelheim Investigational Site 146, Ellhofen
  - Boehringer Ingelheim Investigational Site 147, Emmerich
  - Boehringer Ingelheim Investigational Site 148, Erding
  - Boehringer Ingelheim Investigational Site 149, Erfurt
  - Boehringer Ingelheim Investigational Site 150, Erfurt
  - Boehringer Ingelheim Investigational Site 151, Erfurt
  - Boehringer Ingelheim Investigational Site 152, Erkelenz
  - Boehringer Ingelheim Investigational Site 153, Erkelenz
  - Boehringer Ingelheim Investigational Site 154, Erlangen
  - Boehringer Ingelheim Investigational Site 155, Erlensee
  - Boehringer Ingelheim Investigational Site 156, Eschborn
  - Boehringer Ingelheim Investigational Site 157, Eschwege
  - Boehringer Ingelheim Investigational Site 158, Essen
  - Boehringer Ingelheim Investigational Site 159, Essen
  - Boehringer Ingelheim Investigational Site 160, Essen
  - Boehringer Ingelheim Investigational Site 161, Essen
  - Boehringer Ingelheim Investigational Site 162, Essen
  - Boehringer Ingelheim Investigational Site 163, Essen
  - Boehringer Ingelheim Investigational Site 164, Essen
  - Boehringer Ingelheim Investigational Site 165, Essen
  - Boehringer Ingelheim Investigational Site 166, Essen
  - Boehringer Ingelheim Investigational Site 167, Essen
  - Boehringer Ingelheim Investigational Site 168, Essen
  - Boehringer Ingelheim Investigational Site 169, Essen
  - Boehringer Ingelheim Investigational Site 171, Essen-Werden
  - Boehringer Ingelheim Investigational Site 172, Euskirchen
  - Boehringer Ingelheim Investigational Site 173, Euskirchen
  - Boehringer Ingelheim Investigational Site 174, Eutin
  - Boehringer Ingelheim Investigational Site 175, Eutin
  - Boehringer Ingelheim Investigational Site 176, Eutin
  - Boehringer Ingelheim Investigational Site 177, Falkensee
  - Boehringer Ingelheim Investigational Site 178, Filderstadt
  - Boehringer Ingelheim Investigational Site 179, Finsterwalde
  - Boehringer Ingelheim Investigational Site 180, Flensburg
  - Boehringer Ingelheim Investigational Site 181, Forchheim
  - Boehringer Ingelheim Investigational Site 182, Forchheim
  - Boehringer Ingelheim Investigational Site 183, Forchheim
  - Boehringer Ingelheim Investigational Site 184, Forchheim
  - Boehringer Ingelheim Investigational Site 185, Forchheim
  - Boehringer Ingelheim Investigational Site 186, Framersheim
  - Boehringer Ingelheim Investigational Site 187, Frankfurt
  - Boehringer Ingelheim Investigational Site 188, Frankfurt
  - Boehringer Ingelheim Investigational Site 189, Frankfurt
  - Boehringer Ingelheim Investigational Site 190, Frankfurt
  - Boehringer Ingelheim Investigational Site 191, Frankfurt
  - Boehringer Ingelheim Investigational Site 192, Frankfurt
  - Boehringer Ingelheim Investigational Site 193, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site 194, Freiberg
  - Boehringer Ingelheim Investigational Site 195, Freiberg
  - Boehringer Ingelheim Investigational Site 196, Freising
  - Boehringer Ingelheim Investigational Site 197, Freising
  - Boehringer Ingelheim Investigational Site 198, Freital
  - Boehringer Ingelheim Investigational Site 199, Freital
  - Boehringer Ingelheim Investigational Site 200, Friedrichshafen
  - Boehringer Ingelheim Investigational Site 201, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 202, Friedrichsthal
  - Boehringer Ingelheim Investigational Site 203, Fürstenwalde
  - Boehringer Ingelheim Investigational Site 204, Fürstenwalde
  - Boehringer Ingelheim Investigational Site 205, Fürth
  - Boehringer Ingelheim Investigational Site 206, Gailsdorf
  - Boehringer Ingelheim Investigational Site 207, Gangkofen
  - Boehringer Ingelheim Investigational Site 208, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site 209, Garmisch-Partenkirchen
  - Boehringer Ingelheim Investigational Site 210, Gauting
  - Boehringer Ingelheim Investigational Site 211, Gelnhausen
  - Boehringer Ingelheim Investigational Site 212, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 213, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 214, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 215, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 216, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 217, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 218, Gelsenkirchen
  - Boehringer Ingelheim Investigational Site 219, Geltow
  - Boehringer Ingelheim Investigational Site 220, Geretsried
  - Boehringer Ingelheim Investigational Site 221, Germersheim
  - Boehringer Ingelheim Investigational Site 222, Gevelsberg
  - Boehringer Ingelheim Investigational Site 223, Goslar
  - Boehringer Ingelheim Investigational Site 224, Gräfeling
  - Boehringer Ingelheim Investigational Site 225, Greußen
  - Boehringer Ingelheim Investigational Site 226, Grevesmühlen
  - Boehringer Ingelheim Investigational Site 227, Grimma
  - Boehringer Ingelheim Investigational Site 228, Großrosseln
  - Boehringer Ingelheim Investigational Site 229, Gummersbach
  - Boehringer Ingelheim Investigational Site 230, Gundelfingen
  - Boehringer Ingelheim Investigational Site 231, Gütersloh
  - Boehringer Ingelheim Investigational Site 232, Gütersloh
  - Boehringer Ingelheim Investigational Site 233, Gütersloh
  - Boehringer Ingelheim Investigational Site 234, Gütersloh
  - Boehringer Ingelheim Investigational Site 235, Gütersloh
  - Boehringer Ingelheim Investigational Site 236, Gütersloh
  - Boehringer Ingelheim Investigational Site 237, Hagen
  - Boehringer Ingelheim Investigational Site 238, Hagen
  - Boehringer Ingelheim Investigational Site 239, Hagen
  - Boehringer Ingelheim Investigational Site 240, Halberstadt
  - Boehringer Ingelheim Investigational Site 241, Haldensleben I
  - Boehringer Ingelheim Investigational Site 242, Haldensleben I
  - Boehringer Ingelheim Investigational Site 243, Halle
  - Boehringer Ingelheim Investigational Site 244, Halle
  - Boehringer Ingelheim Investigational Site 245, Halle
  - Boehringer Ingelheim Investigational Site 246, Halle
  - Boehringer Ingelheim Investigational Site 247, Halle
  - Boehringer Ingelheim Investigational Site 248, Halle
  - Boehringer Ingelheim Investigational Site 249, Halle
  - Boehringer Ingelheim Investigational Site 250, Hallstadt
  - Boehringer Ingelheim Investigational Site 251, Hamburg
  - Boehringer Ingelheim Investigational Site 252, Hamburg
  - Boehringer Ingelheim Investigational Site 253, Hamburg
  - Boehringer Ingelheim Investigational Site 254, Hamburg
  - Boehringer Ingelheim Investigational Site 255, Hamburg
  - Boehringer Ingelheim Investigational Site 256, Hamburg
  - Boehringer Ingelheim Investigational Site 257, Hamburg
  - Boehringer Ingelheim Investigational Site 258, Hamburg
  - Boehringer Ingelheim Investigational Site 259, Hamburg
  - Boehringer Ingelheim Investigational Site 260, Hamburg
  - Boehringer Ingelheim Investigational Site 261, Hamelin
  - Boehringer Ingelheim Investigational Site 262, Hanerau-Hademarschen
  - Boehringer Ingelheim Investigational Site 263, Hanover
  - Boehringer Ingelheim Investigational Site 264, Hanover
  - Boehringer Ingelheim Investigational Site 265, Hanover
  - Boehringer Ingelheim Investigational Site 266, Hanover
  - Boehringer Ingelheim Investigational Site 267, Hartha
  - Boehringer Ingelheim Investigational Site 268, Hartha
  - Boehringer Ingelheim Investigational Site 269, Heide
  - Boehringer Ingelheim Investigational Site 270, Heidelberg
  - Boehringer Ingelheim Investigational Site 271, Heidelberg
  - Boehringer Ingelheim Investigational Site 272, Heidelberg
  - Boehringer Ingelheim Investigational Site 273, Heidelberg
  - Boehringer Ingelheim Investigational Site 274, Heidelberg
  - Boehringer Ingelheim Investigational Site 275, Heilbronn
  - Boehringer Ingelheim Investigational Site 276, Heilbronn
  - Boehringer Ingelheim Investigational Site 277, Heilbronn
  - Boehringer Ingelheim Investigational Site 278, Heilbronn
  - Boehringer Ingelheim Investigational Site 279, Heilbronn
  - Boehringer Ingelheim Investigational Site 280, Heinsberg-Karken
  - Boehringer Ingelheim Investigational Site 281, Hellenthal
  - Boehringer Ingelheim Investigational Site 62, Hellersdorf
  - Boehringer Ingelheim Investigational Site 63, Hellersdorf
  - Boehringer Ingelheim Investigational Site 282, Helmstedt
  - Boehringer Ingelheim Investigational Site 283, Hemmingen
  - Boehringer Ingelheim Investigational Site 284, Hemmingen
  - Boehringer Ingelheim Investigational Site 285, Hemmingen
  - Boehringer Ingelheim Investigational Site 286, Hemmingen
  - Boehringer Ingelheim Investigational Site 287, Hemsbach
  - Boehringer Ingelheim Investigational Site 288, Hemsbach
  - Boehringer Ingelheim Investigational Site 289, Herbsleben
  - Boehringer Ingelheim Investigational Site 290, Herford
  - Boehringer Ingelheim Investigational Site 291, Herne
  - Boehringer Ingelheim Investigational Site 292, Herne
  - Boehringer Ingelheim Investigational Site 293, Herne
  - Boehringer Ingelheim Investigational Site 294, Hettstedt
  - Boehringer Ingelheim Investigational Site 295, Hilden
  - Boehringer Ingelheim Investigational Site 296, Hilden
  - Boehringer Ingelheim Investigational Site 297, Hildesheim
  - Boehringer Ingelheim Investigational Site 298, Hirschau
  - Boehringer Ingelheim Investigational Site 299, Hohenau
  - Boehringer Ingelheim Investigational Site 300, Homburg
  - Boehringer Ingelheim Investigational Site 301, Homburg/Saar
  - Boehringer Ingelheim Investigational Site 302, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 303, Hoyerswerda
  - Boehringer Ingelheim Investigational Site 307, Hummeltal
  - Boehringer Ingelheim Investigational Site 304, Hückelhoven
  - Boehringer Ingelheim Investigational Site 305, Hückelhoven
  - Boehringer Ingelheim Investigational Site 306, Hüffenhardt
  - Boehringer Ingelheim Investigational Site 308, Ibbenbueren
  - Boehringer Ingelheim Investigational Site 309, Irsch/Saar
  - Boehringer Ingelheim Investigational Site 310, Issum
  - Boehringer Ingelheim Investigational Site 311, Issum
  - Boehringer Ingelheim Investigational Site 312, Jena
  - Boehringer Ingelheim Investigational Site 313, Jena
  - Boehringer Ingelheim Investigational Site 314, Jerichow
  - Boehringer Ingelheim Investigational Site 315, Jessen
  - Boehringer Ingelheim Investigational Site 316, Kaiserslautern
  - Boehringer Ingelheim Investigational Site 99, Kalawa
  - Boehringer Ingelheim Investigational Site 317, Kalkar
  - Boehringer Ingelheim Investigational Site 318, Kamen
  - Boehringer Ingelheim Investigational Site 319, Karlsruhe
  - Boehringer Ingelheim Investigational Site 320, Karlsruhe
  - Boehringer Ingelheim Investigational Site 321, Kassel
  - Boehringer Ingelheim Investigational Site 322, Katzenelnbogen
  - Boehringer Ingelheim Investigational Site 323, Kempen
  - Boehringer Ingelheim Investigational Site 170, Kettwig
  - Boehringer Ingelheim Investigational Site 324, Kevelaer
  - Boehringer Ingelheim Investigational Site 325, Kiel
  - Boehringer Ingelheim Investigational Site 326, Kierspe
  - Boehringer Ingelheim Investigational Site 327, Kirchenlamitz
  - Boehringer Ingelheim Investigational Site 328, Kirchheilingen
  - Boehringer Ingelheim Investigational Site 329, Kirchheim/Teck
  - Boehringer Ingelheim Investigational Site 330, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site 331, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site 332, Kirchheimbolanden
  - Boehringer Ingelheim Investigational Site 333, Kitzingen
  - Boehringer Ingelheim Investigational Site 334, Kleinmachnow
  - Boehringer Ingelheim Investigational Site 335, Kleinmachnow
  - Boehringer Ingelheim Investigational Site 336, Koblenz
  - Boehringer Ingelheim Investigational Site 337, Koblenz
  - Boehringer Ingelheim Investigational Site 338, Koblenz
  - Boehringer Ingelheim Investigational Site 339, Koblenz
  - Boehringer Ingelheim Investigational Site 354, Köln-Lindenthal
  - Boehringer Ingelheim Investigational Site 355, Köthen
  - Boehringer Ingelheim Investigational Site 356, Krefeld
  - Boehringer Ingelheim Investigational Site 357, Krefeld
  - Boehringer Ingelheim Investigational Site 358, Krefeld
  - Boehringer Ingelheim Investigational Site 359, Krefeld
  - Boehringer Ingelheim Investigational Site 360, Krefeld
  - Boehringer Ingelheim Investigational Site 361, Krumbach
  - Boehringer Ingelheim Investigational Site 362, Künzing
  - Boehringer Ingelheim Investigational Site 363, Künzing
  - Boehringer Ingelheim Investigational Site 364, Kyritz
  - Boehringer Ingelheim Investigational Site 365, Laaber
  - Boehringer Ingelheim Investigational Site 366, Lahnau
  - Boehringer Ingelheim Investigational Site 367, Landshut
  - Boehringer Ingelheim Investigational Site 368, Landshut
  - Boehringer Ingelheim Investigational Site 369, Landstuhl
  - Boehringer Ingelheim Investigational Site 370, Langen
  - Boehringer Ingelheim Investigational Site 371, Langenfeld
  - Boehringer Ingelheim Investigational Site 372, Lauenburg
  - Boehringer Ingelheim Investigational Site 373, Lauenburg
  - Boehringer Ingelheim Investigational Site 374, Leiblfing
  - Boehringer Ingelheim Investigational Site 375, Leipzig
  - Boehringer Ingelheim Investigational Site 376, Leipzig
  - Boehringer Ingelheim Investigational Site 377, Leipzig
  - Boehringer Ingelheim Investigational Site 378, Leipzig
  - Boehringer Ingelheim Investigational Site 379, Leipzig
  - Boehringer Ingelheim Investigational Site 380, Leipzig
  - Boehringer Ingelheim Investigational Site 381, Leipzig
  - Boehringer Ingelheim Investigational Site 382, Leipzig
  - Boehringer Ingelheim Investigational Site 383, Leipzig
  - Boehringer Ingelheim Investigational Site 384, Leipzig
  - Boehringer Ingelheim Investigational Site 385, Leonberg
  - Boehringer Ingelheim Investigational Site 386, Leverkusen
  - Boehringer Ingelheim Investigational Site 387, Leverkusen
  - Boehringer Ingelheim Investigational Site 388, Leverkusen
  - Boehringer Ingelheim Investigational Site 389, Leverkusen
  - Boehringer Ingelheim Investigational Site 390, Lichtenfels
  - Boehringer Ingelheim Investigational Site 391, Lichtenfels
  - Boehringer Ingelheim Investigational Site 392, Limburgerhof
  - Boehringer Ingelheim Investigational Site 395, Luckenwalde
  - Boehringer Ingelheim Investigational Site 396, Luckenwalde
  - Boehringer Ingelheim Investigational Site 400, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 401, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 402, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 403, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 404, Ludwigshafen
  - Boehringer Ingelheim Investigational Site 393, Lübeck
  - Boehringer Ingelheim Investigational Site 397, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 398, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 399, Lüdenscheid
  - Boehringer Ingelheim Investigational Site 405, Machern
  - Boehringer Ingelheim Investigational Site 406, Magdeburg
  - Boehringer Ingelheim Investigational Site 407, Magdeburg
  - Boehringer Ingelheim Investigational Site 408, Magdeburg
  - Boehringer Ingelheim Investigational Site 409, Mainz
  - Boehringer Ingelheim Investigational Site 410, Mannheim
  - Boehringer Ingelheim Investigational Site 411, Mannheim
  - Boehringer Ingelheim Investigational Site 412, Mannheim
  - Boehringer Ingelheim Investigational Site 413, Mannheim
  - Boehringer Ingelheim Investigational Site 414, Mannheim
  - Boehringer Ingelheim Investigational Site 415, Mannheim - Vogelstang
  - Boehringer Ingelheim Investigational Site 416, Marburg
  - Boehringer Ingelheim Investigational Site 417, Marburg
  - Boehringer Ingelheim Investigational Site 418, Marburg
  - Boehringer Ingelheim Investigational Site 419, Marktleugast
  - Boehringer Ingelheim Investigational Site 420, Marktredwitz
  - Boehringer Ingelheim Investigational Site 421, Marl
  - Boehringer Ingelheim Investigational Site 422, Meckenheim
  - Boehringer Ingelheim Investigational Site 423, Meckenheim
  - Boehringer Ingelheim Investigational Site 424, Meeder
  - Boehringer Ingelheim Investigational Site 425, Meinerzhagen
  - Boehringer Ingelheim Investigational Site 426, Menden
  - Boehringer Ingelheim Investigational Site 427, Menden
  - Boehringer Ingelheim Investigational Site 428, Menden
  - Boehringer Ingelheim Investigational Site 429, Menden
  - Boehringer Ingelheim Investigational Site 430, Michelstadt
  - Boehringer Ingelheim Investigational Site 431, Minden
  - Boehringer Ingelheim Investigational Site 432, Minden
  - Boehringer Ingelheim Investigational Site 433, Minden
  - Boehringer Ingelheim Investigational Site 434, Moers
  - Boehringer Ingelheim Investigational Site 435, Molfsee
  - Boehringer Ingelheim Investigational Site 438, Monheim
  - Boehringer Ingelheim Investigational Site 439, Moosinning
  - Boehringer Ingelheim Investigational Site 440, Morbach
  - Boehringer Ingelheim Investigational Site 436, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 437, Mönchengladbach
  - Boehringer Ingelheim Investigational Site 441, Mühldorf/Inn
  - Boehringer Ingelheim Investigational Site 442, Mühlmein Am Main - Lämmerspiel
  - Boehringer Ingelheim Investigational Site 443, Mülheim
  - Boehringer Ingelheim Investigational Site 444, Mülheim
  - Boehringer Ingelheim Investigational Site 445, Mülsen
  - Boehringer Ingelheim Investigational Site 446, München
  - Boehringer Ingelheim Investigational Site 447, München
  - Boehringer Ingelheim Investigational Site 448, München
  - Boehringer Ingelheim Investigational Site 449, München
  - Boehringer Ingelheim Investigational Site 450, München
  - Boehringer Ingelheim Investigational Site 451, München
  - Boehringer Ingelheim Investigational Site 452, München
  - Boehringer Ingelheim Investigational Site 453, Münnerstadt
  - Boehringer Ingelheim Investigational Site 454, Münnerstadt
  - Boehringer Ingelheim Investigational Site 455, Münnerstadt
  - Boehringer Ingelheim Investigational Site 457, Münster
  - Boehringer Ingelheim Investigational Site 458, Münster
  - Boehringer Ingelheim Investigational Site 459, Naumburg
  - Boehringer Ingelheim Investigational Site 462, Neu-Isenburg
  - Boehringer Ingelheim Investigational Site 460, Neuburg an der Donau
  - Boehringer Ingelheim Investigational Site 461, Neufahrn
  - Boehringer Ingelheim Investigational Site 463, Neukirchen
  - Boehringer Ingelheim Investigational Site 464, Neumarkt
  - Boehringer Ingelheim Investigational Site 465, Neumarkt
  - Boehringer Ingelheim Investigational Site 466, Neuss
  - Boehringer Ingelheim Investigational Site 467, Neustadt
  - Boehringer Ingelheim Investigational Site 468, Neuwied
  - Boehringer Ingelheim Investigational Site 469, Niederwörresbach
  - Boehringer Ingelheim Investigational Site 470, Nienburg
  - Boehringer Ingelheim Investigational Site 471, Nienburg
  - Boehringer Ingelheim Investigational Site 472, Nienburg
  - Boehringer Ingelheim Investigational Site 473, Niesky
  - Boehringer Ingelheim Investigational Site 474, Nordhausen
  - Boehringer Ingelheim Investigational Site 475, Northeim
  - Boehringer Ingelheim Investigational Site 476, Northeim
  - Boehringer Ingelheim Investigational Site 477, Nuremberg
  - Boehringer Ingelheim Investigational Site 478, Nuremberg
  - Boehringer Ingelheim Investigational Site 479, Nuremberg
  - Boehringer Ingelheim Investigational Site 480, Nuremberg
  - Boehringer Ingelheim Investigational Site 481, Nuremberg
  - Boehringer Ingelheim Investigational Site 482, Nuremberg
  - Boehringer Ingelheim Investigational Site 483, Nuremberg
  - Boehringer Ingelheim Investigational Site 484, Nuremberg
  - Boehringer Ingelheim Investigational Site 485, Nuremberg
  - Boehringer Ingelheim Investigational Site 486, Nuremberg
  - Boehringer Ingelheim Investigational Site 487, Nuremberg
  - Boehringer Ingelheim Investigational Site 488, Nuremberg
  - Boehringer Ingelheim Investigational Site 489, Oberdorla
  - Boehringer Ingelheim Investigational Site 490, Oberhausen
  - Boehringer Ingelheim Investigational Site 491, Oberhausen
  - Boehringer Ingelheim Investigational Site 492, Oberhausen
  - Boehringer Ingelheim Investigational Site 493, Offenbach
  - Boehringer Ingelheim Investigational Site 494, Offenburg
  - Boehringer Ingelheim Investigational Site 495, Oldenburg
  - Boehringer Ingelheim Investigational Site 496, Oranienburg
  - Boehringer Ingelheim Investigational Site 497, Oranienburg
  - Boehringer Ingelheim Investigational Site 498, Oschatz
  - Boehringer Ingelheim Investigational Site 499, Oschersleben
  - Boehringer Ingelheim Investigational Site 500, Osterode
  - Boehringer Ingelheim Investigational Site 501, Ostrach
  - Boehringer Ingelheim Investigational Site 502, Ostrach
  - Boehringer Ingelheim Investigational Site 503, Papenburg
  - Boehringer Ingelheim Investigational Site 504, Papenburg
  - Boehringer Ingelheim Investigational Site 505, Papenburg
  - Boehringer Ingelheim Investigational Site 506, Passau
  - Boehringer Ingelheim Investigational Site 507, Petersberg
  - Boehringer Ingelheim Investigational Site 508, Plauen
  - Boehringer Ingelheim Investigational Site 509, Potsdam
  - Boehringer Ingelheim Investigational Site 510, Potsdam
  - Boehringer Ingelheim Investigational Site 511, Potsdam
  - Boehringer Ingelheim Investigational Site 512, Potsdam
  - Boehringer Ingelheim Investigational Site 513, Potsdam
  - Boehringer Ingelheim Investigational Site 514, Potsdam
  - Boehringer Ingelheim Investigational Site 515, Potsdam
  - Boehringer Ingelheim Investigational Site 516, Preetz
  - Boehringer Ingelheim Investigational Site 517, Pullach
  - Boehringer Ingelheim Investigational Site 518, Radebeul
  - Boehringer Ingelheim Investigational Site 519, Radebeul
  - Boehringer Ingelheim Investigational Site 520, Radebeul
  - Boehringer Ingelheim Investigational Site 521, Radebeul
  - Boehringer Ingelheim Investigational Site 522, Radebeul
  - Boehringer Ingelheim Investigational Site 523, Radebeul
  - Boehringer Ingelheim Investigational Site 524, Radebeul
  - Boehringer Ingelheim Investigational Site 525, Radebeul
  - Boehringer Ingelheim Investigational Site 526, Rathenow
  - Boehringer Ingelheim Investigational Site 527, Ratingen
  - Boehringer Ingelheim Investigational Site 528, Ratingen
  - Boehringer Ingelheim Investigational Site 529, Raubach
  - Boehringer Ingelheim Investigational Site 530, Ravensburg
  - Boehringer Ingelheim Investigational Site 531, Rehau
  - Boehringer Ingelheim Investigational Site 532, Rellingen
  - Boehringer Ingelheim Investigational Site 533, Remscheid
  - Boehringer Ingelheim Investigational Site 534, Remscheid
  - Boehringer Ingelheim Investigational Site 535, Remscheid
  - Boehringer Ingelheim Investigational Site 536, Rendsburg
  - Boehringer Ingelheim Investigational Site 537, Rheinfelden
  - Boehringer Ingelheim Investigational Site 538, Rickenbach
  - Boehringer Ingelheim Investigational Site 539, Riedstadt
  - Boehringer Ingelheim Investigational Site 540, Rodalben
  - Boehringer Ingelheim Investigational Site 541, Rodalben
  - Boehringer Ingelheim Investigational Site 542, Rostock
  - Boehringer Ingelheim Investigational Site 543, Rostock
  - Boehringer Ingelheim Investigational Site 544, Rostock
  - Boehringer Ingelheim Investigational Site 545, Rostock
  - Boehringer Ingelheim Investigational Site 546, Rostock
  - Boehringer Ingelheim Investigational Site 547, Roth
  - Boehringer Ingelheim Investigational Site 548, Roth
  - Boehringer Ingelheim Investigational Site 549, Rüdersdorf
  - Boehringer Ingelheim Investigational Site 550, Rüdersdorf
  - Boehringer Ingelheim Investigational Site 551, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 552, Rüsselsheim am Main
  - Boehringer Ingelheim Investigational Site 553, Saalfeld
  - Boehringer Ingelheim Investigational Site 554, Saarbrücken
  - Boehringer Ingelheim Investigational Site 555, Saarbrücken
  - Boehringer Ingelheim Investigational Site 556, Saarbrücken
  - Boehringer Ingelheim Investigational Site 557, Saarbrücken
  - Boehringer Ingelheim Investigational Site 558, Saarbrücken
  - Boehringer Ingelheim Investigational Site 559, Saarbrücken
  - Boehringer Ingelheim Investigational Site 560, Saarlouis
  - Boehringer Ingelheim Investigational Site 561, Saarlouis
  - Boehringer Ingelheim Investigational Site 562, Saarlouis
  - Boehringer Ingelheim Investigational Site 563, Saarlouis
  - Boehringer Ingelheim Investigational Site 564, Saarlouis
  - Boehringer Ingelheim Investigational Site 565, Saarlouis
  - Boehringer Ingelheim Investigational Site 566, Saarlouis
  - Boehringer Ingelheim Investigational Site 567, Sand
  - Boehringer Ingelheim Investigational Site 568, Schenefeld
  - Boehringer Ingelheim Investigational Site 569, Schleswig
  - Boehringer Ingelheim Investigational Site 570, Schleswig
  - Boehringer Ingelheim Investigational Site 571, Schmölln
  - Boehringer Ingelheim Investigational Site 572, Schmölln
  - Boehringer Ingelheim Investigational Site 573, Schmölln
  - Boehringer Ingelheim Investigational Site 574, Schönsee
  - Boehringer Ingelheim Investigational Site 575, Schwandorf in Bayern
  - Boehringer Ingelheim Investigational Site 576, Schwedt
  - Boehringer Ingelheim Investigational Site 577, Schwerin
  - Boehringer Ingelheim Investigational Site 578, Schwerin
  - Boehringer Ingelheim Investigational Site 579, Schwetzingen
  - Boehringer Ingelheim Investigational Site 580, Sebnitz
  - Boehringer Ingelheim Investigational Site 581, Selm
  - Boehringer Ingelheim Investigational Site 582, Sendenhorst
  - Boehringer Ingelheim Investigational Site 583, Siegen
  - Boehringer Ingelheim Investigational Site 584, Siegen
  - Boehringer Ingelheim Investigational Site 585, Simmern
  - Boehringer Ingelheim Investigational Site 586, Simmertal
  - Boehringer Ingelheim Investigational Site 587, Sinsheim
  - Boehringer Ingelheim Investigational Site 588, Sobernheim
  - Boehringer Ingelheim Investigational Site 589, Soltau
  - Boehringer Ingelheim Investigational Site 590, Sondershausen
  - Boehringer Ingelheim Investigational Site 591, Sonsbeck
  - Boehringer Ingelheim Investigational Site 592, Sprendlingen
  - Boehringer Ingelheim Investigational Site 593, Stade
  - Boehringer Ingelheim Investigational Site 594, Stadland-Schwei
  - Boehringer Ingelheim Investigational Site 595, Starnberg
  - Boehringer Ingelheim Investigational Site 596, Staudernheim
  - Boehringer Ingelheim Investigational Site 597, Steinbach
  - Boehringer Ingelheim Investigational Site 598, Steinfurt
  - Boehringer Ingelheim Investigational Site 599, Steinhagen
  - Boehringer Ingelheim Investigational Site 600, Steinhagen
  - Boehringer Ingelheim Investigational Site 601, Steinhagen
  - Boehringer Ingelheim Investigational Site 602, Steinhagen
  - Boehringer Ingelheim Investigational Site 603, Steinhagen
  - Boehringer Ingelheim Investigational Site 604, Steinhagen
  - Boehringer Ingelheim Investigational Site 605, Stockach
  - Boehringer Ingelheim Investigational Site 606, Stödtlen
  - Boehringer Ingelheim Investigational Site 607, Straubing
  - Boehringer Ingelheim Investigational Site 608, Strausberg
  - Boehringer Ingelheim Investigational Site 609, Stuttgart
  - Boehringer Ingelheim Investigational Site 610, Stuttgart
  - Boehringer Ingelheim Investigational Site 611, Stuttgart
  - Boehringer Ingelheim Investigational Site 612, Stuttgart
  - Boehringer Ingelheim Investigational Site 613, Stuttgart
  - Boehringer Ingelheim Investigational Site 614, Sünna
  - Boehringer Ingelheim Investigational Site 615, Süßen
  - Boehringer Ingelheim Investigational Site 616, Teltow
  - Boehringer Ingelheim Investigational Site 617, Teterow
  - Boehringer Ingelheim Investigational Site 618, Teuchern
  - Boehringer Ingelheim Investigational Site 619, Teuchern
  - Boehringer Ingelheim Investigational Site 621, Titisee-Neustadt
  - Boehringer Ingelheim Investigational Site 622, Töging
  - Boehringer Ingelheim Investigational Site 623, Tönisvorst
  - Boehringer Ingelheim Investigational Site 624, Tönisvorst
  - Boehringer Ingelheim Investigational Site 394, Travemünde
  - Boehringer Ingelheim Investigational Site 625, Troisdorf
  - Boehringer Ingelheim Investigational Site 626, Tüßling
  - Boehringer Ingelheim Investigational Site 627, Uchte
  - Boehringer Ingelheim Investigational Site 628, Ulm
  - Boehringer Ingelheim Investigational Site 629, Ulm
  - Boehringer Ingelheim Investigational Site 630, Ulm
  - Boehringer Ingelheim Investigational Site 631, Ulm
  - Boehringer Ingelheim Investigational Site 632, Ulm
  - Boehringer Ingelheim Investigational Site 633, Ulm
  - Boehringer Ingelheim Investigational Site 634, Ulm
  - Boehringer Ingelheim Investigational Site 635, Undenheim
  - Boehringer Ingelheim Investigational Site 636, Unterschneidheim
  - Boehringer Ingelheim Investigational Site 637, Uttenreuth
  - Boehringer Ingelheim Investigational Site 638, Uttenreuth
  - Boehringer Ingelheim Investigational Site 639, Veringenstadt
  - Boehringer Ingelheim Investigational Site 640, Veringenstadt
  - Boehringer Ingelheim Investigational Site 641, Villingen-Schwenningen
  - Boehringer Ingelheim Investigational Site 642, Visselhövede
  - Boehringer Ingelheim Investigational Site 643, Völklingen
  - Boehringer Ingelheim Investigational Site 644, Wachenheim
  - Boehringer Ingelheim Investigational Site 645, Waren
  - Boehringer Ingelheim Investigational Site 646, Warendorf
  - Boehringer Ingelheim Investigational Site 647, Warendorf
  - Boehringer Ingelheim Investigational Site 648, Warendorf
  - Boehringer Ingelheim Investigational Site 649, Warendorf
  - Boehringer Ingelheim Investigational Site 650, Warendorf
  - Boehringer Ingelheim Investigational Site 651, Warendorf
  - Boehringer Ingelheim Investigational Site 652, Warthausen
  - Boehringer Ingelheim Investigational Site 653, Wegberg
  - Boehringer Ingelheim Investigational Site 654, Wehrheim
  - Boehringer Ingelheim Investigational Site 655, Weißenhorn
  - Boehringer Ingelheim Investigational Site 656, Wertheim am Main
  - Boehringer Ingelheim Investigational Site 657, Westerburg
  - Boehringer Ingelheim Investigational Site 658, Wettenberg
  - Boehringer Ingelheim Investigational Site 659, Wetzlar
  - Boehringer Ingelheim Investigational Site 660, Wetzlar
  - Boehringer Ingelheim Investigational Site 661, Wetzlar
  - Boehringer Ingelheim Investigational Site 662, Wiesbaden
  - Boehringer Ingelheim Investigational Site 663, Wiesbaden
  - Boehringer Ingelheim Investigational Site 664, Wiesbaden
  - Boehringer Ingelheim Investigational Site 665, Wiesbaden
  - Boehringer Ingelheim Investigational Site 666, Wiesbaden
  - Boehringer Ingelheim Investigational Site 667, Wiesbaden
  - Boehringer Ingelheim Investigational Site 668, Wiesbaden
  - Boehringer Ingelheim Investigational Site 669, Wiesbaden
  - Boehringer Ingelheim Investigational Site 670, Wiesbaden
  - Boehringer Ingelheim Investigational Site 671, Wiesbaden
  - Boehringer Ingelheim Investigational Site 672, Wiesbaden
  - Boehringer Ingelheim Investigational Site 673, Wiesbaden
  - Boehringer Ingelheim Investigational Site 674, Wiesloch
  - Boehringer Ingelheim Investigational Site 675, Wiesloch
  - Boehringer Ingelheim Investigational Site 676, Wiesloch
  - Boehringer Ingelheim Investigational Site 677, Wiesloch
  - Boehringer Ingelheim Investigational Site 678, Wiesloch
  - Boehringer Ingelheim Investigational Site 679, Wiesloch
  - Boehringer Ingelheim Investigational Site 680, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 681, Wilhelmshaven
  - Boehringer Ingelheim Investigational Site 682, Willich
  - Boehringer Ingelheim Investigational Site 683, Winhönng
  - Boehringer Ingelheim Investigational Site 684, Witten
  - Boehringer Ingelheim Investigational Site 685, Witten
  - Boehringer Ingelheim Investigational Site 686, Witten
  - Boehringer Ingelheim Investigational Site 687, Witten
  - Boehringer Ingelheim Investigational Site 688, Wittenberg
  - Boehringer Ingelheim Investigational Site 689, Wittenberg
  - Boehringer Ingelheim Investigational Site 690, Wolfenbüttel
  - Boehringer Ingelheim Investigational Site 691, Wolfsburg
  - Boehringer Ingelheim Investigational Site 692, Wolfsburg
  - Boehringer Ingelheim Investigational Site 693, Wolfsburg
  - Boehringer Ingelheim Investigational Site 694, Wolfsburg
  - Boehringer Ingelheim Investigational Site 695, Wolfsburg - Fallersleben
  - Boehringer Ingelheim Investigational Site 696, Wörth
  - Boehringer Ingelheim Investigational Site 697, Wörth
  - Boehringer Ingelheim Investigational Site 698, Wuppertal
  - Boehringer Ingelheim Investigational Site 699, Zellertal
  - Boehringer Ingelheim Investigational Site 700, Zerbst
  - Boehringer Ingelheim Investigational Site 701, Zirndorf
  - Boehringer Ingelheim Investigational Site 702, Zirndorf
  - Boehringer Ingelheim Investigational Site 703, Zweibrücken

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open, prospective non-interventional study in patients with moderate to severe chronic obstructive pulmonary disease (COPD).
Groups:
- All Patients: Patients with moderate to severe chronic obstructive pulmonary disease (COPD) and treated with Spiriva Respimat plus Striverdi Respimat or Spiriva 18 microgram plus Striverdi Respimat
Period: Overall Study
Arm/Group | All Patients
Started | 1858
Completed | 1854
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: Treated set which includes all patients with baseline visit data.
Arm/Group | All Patients
Number analyzed (Participants) | 1858
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.41 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 770
  Male | 1088

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With "Therapeutic Success"
Description: Percentage of participants with "therapeutic success" defined as a 10-point increase in the physical activity assessed by patient´s questionnaire (PF-10) score between the initial examination and after 4-6 weeks.
  The PF-10 score is a subscale of the quality of life questionnaire Short Form 36 (SF-36) and contains 10 questions concerning physical activity and capacity. The total score ranges from 0 to 100. A higher score indicates a better physical functioning.
Time Frame: Baseline and 4-6 weeks
Population: Full analysis (FAS) which includes all patients enrolled in the study who did not violated any inclusion or exclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1726
Percentage of participants
  Therapy successful | 48.90
  Therapy not successful | 51.10

2. Secondary Outcome: Absolute Changes in the PF-10 Score
Description: Absolute changes in the PF-10 score.
  The PF-10 score is a subscale of the quality of life questionnaire Short Form 36 (SF-36) and contains 10 questions concerning physical activity and capacity. The total score ranges from 0 to 100. A higher score indicates a better physical functioning.
Time Frame: 4-6 weeks
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Patients
Number analyzed (Participants) | 1726
Units on a scale | 10.15 (19.22)

3. Secondary Outcome: General Health of the Patient at Baseline
Description: General health of the patient as evaluated by the physician using the Physician´s Global Evaluation (PGE) score at the initial examination.
  The PGE score consists of an 8-point-scale which extends from 1 (very bad) to 8 (excellent).
Time Frame: Baseline
Population: FAS including patients with available PGE score at baseline
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1853
Percentage of participants
  1 (poor) | 2.10
  2 | 14.72
  3 | 25.73
  4 | 29.13
  5 | 16.57
  6 | 9.44
  7 | 2.16
  8 (excellent) | 0.11

4. Secondary Outcome: General Health of the Patient After 4-6 Weeks
Description: General health of the patient as evaluated by the physician using the Physician´s Global Evaluation (PGE) score after 4-6 weeks.
  The PGE score consists of an 8-point-scale which extends from 1 (very bad) to 8 (excellent).
Time Frame: 4-6 weeks
Population: FAS including patients with available PGE score at end of study visit
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1770
Percentage of participants
  1 (poor) | 0.96
  2 | 5.48
  3 | 13.67
  4 | 22.60
  5 | 25.08
  6 | 22.09
  7 | 8.25
  8 (excellent) | 1.86

5. Secondary Outcome: Patient Satisfaction: Overall Satisfaction
Description: Patient satisfaction with Spiriva Respimat plus Striverdi Respimat or Spiriva 18 Microgram plus Striverdi Respimat.
  Patient´s satisfaction with study treatment and handling of the Respimat inhaler was assessed on a 7-point-ordinal scale extending from very satisfied (1) to very unsatisfied (7).
Time Frame: 4-6 weeks
Population: FAS including patients with available satisfaction data
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1773
Percentage of participants
  Very satisifed | 25.21
  Satisfied | 42.13
  Rather satisfied | 13.53
  Neither satisfied or dissatisfied | 9.70
  Rather dissatisfied | 4.29
  Dissatisfied | 4.06
  Very dissatisfied | 1.07

6. Secondary Outcome: Patient Satisfaction: Satisfaction With Inhaler
Description: as for outcome 5
Time Frame: 4-6 weeks
Population: FAS including patients with available inhaler satisfaction data
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1779
Percentage of participants
  Very satisifed | 31.53
  Satisfied | 49.86
  Rather satisfied | 10.06
  Neither satisfied or dissatisfied | 5.12
  Rather dissatisfied | 1.52
  Dissatisfied | 1.46
  Very dissatisfied | 0.45

7. Secondary Outcome: Patient Satisfaction: Satisfaction With Handling of Inhaler
Description: as for outcome 5
Time Frame: 4-6 weeks
Population: FAS including patients with available handling of inhaler satisfaction data
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 1778
Percentage of participants
  Very satisifed | 31.44
  Satisfied | 49.32
  Rather satisfied | 11.25
  Neither satisfied or dissatisfied | 5.06
  Rather dissatisfied | 1.57
  Dissatisfied | 0.96
  Very dissatisfied | 0.39

ADVERSE EVENTS:
Time Frame: From start of study until 21 days after permanent discontinuation of study therapy or end of study, up to 9 weeks
Groups:
- Spiriva Respimat + Striverdi Respimat: Patients with moderate to severe chronic obstructive pulmonary disease (COPD) and treated with Spiriva Respimat plus Striverdi Respimat
- Spiriva 18 mcg + Striverdi Respimat: Patients with moderate to severe chronic obstructive pulmonary disease (COPD) and treated with Spiriva 18 microgram plus Striverdi Respimat
Arm/Group | Spiriva Respimat + Striverdi Respimat | Spiriva 18 mcg + Striverdi Respimat
Serious Adverse Events (participants affected / at risk) | 30/1298 | 12/560
Other Adverse Events (participants affected / at risk) | 0/1298 | 0/560
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Spiriva Respimat + Striverdi Respimat (N=1298) | Spiriva 18 mcg + Striverdi Respimat (N=560)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 1
Sudden cardiac death (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gingivitis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes